CLINICAL TRIAL: NCT06925087
Title: Myofascial Release Versus Kinesio Taping: Which is More Effective for Dysmenorrhea Relief
Brief Title: Comparison of Acute Effects of Myofascial Release and Kinesio Taping® in Dysmenorrhea
Acronym: Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Mehmet Miçooğulları, Asst. Prof. Dr., Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0037
Record Dates: First submitted 2025-04-06; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Kinesio Taping; Myofascial Release Technique; Pain; Primary Dysmenorrhea (PD)
Keywords: Kinesio Taping; Menstruation; Primary dysmenorrhea; Myofascial release technique; Physiotherapy
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All treatments will be performed by the same physiotherapist, and assessments will be conducted twice: pre-treatment and post-treatment. Post-treatment assessments will be performed after the third MRT session for Group 1 and 72 hours after the KT application for Group 2. This will be a single-blind study, with all assessments carried out by a physiotherapist blinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Release Technique Group (Active Comparator): During the application of Myofascial Release Technique (MRT), the fingers or hand will be first placed on the treatment area. Pressure will be applied to the soft tissue until the restricted layer was felt, and then the fascia was moved along the surface of the underlying layers while maintaining contact with the deeper layers. Tension will be applied for approximately 60-90 seconds, and if a release will not felt, the duration will extended until the release occurred. MRT will be performed with dry hands, without the use of any intermediary substances, and will be applied in both supine and prone positions. In the treatment program, anterolateral release techniques (targeting fascia superficialis, fascia transversalis, and fascia extraperitonealis) will be applied in the supine position, while posterior release techniques (targeting fascia thoracolumbalis and erector spinae) will be applied in the prone position.
  Interventions: Other: Myofascial Release Technique
- Kinesio Taping Group (Active Comparator): Two different techniques will be used in the Kinesio Taping application. First, four I-shaped Kinesio tapes (Kinesio Tex® Gold), each 5 cm wide and 0.5 mm thick, will be applied in a star-shaped pattern using the "space correction technique" with 25-50% tension at the S2-S4 level (sacral region) while the participant will in a seated position. Additionally, to direct the uterus into retroversion during menstruation, a 15 cm long I-shaped tape will be applied to the suprapubic region using the "ligament correction technique" with 100% tension.
  Interventions: Other: Kinesio Taping Technique
- Control Group (No Intervention): No intervention will be applied to the control group. After the study will be completed, participants in the control group will be offered their preferred treatment option.

INTERVENTIONS:
Other: Myofascial Release Technique — During the application of Myofascial Release Technique (MRT), the fingers or hand will be first placed on the treatment area. Pressure will be applied to the soft tissue until the restricted layer was felt, and then the fascia was moved along the surface of the underlying layers while maintaining contact with the deeper layers. Tension will be applied for approximately 60-90 seconds, and if a release will not felt, the duration will extended until the release occurred. MRT will be performed with dry hands, without the use of any intermediary substances, and will be applied in both supine and prone positions. In the treatment program, anterolateral release techniques (targeting fascia superficialis, fascia transversalis, and fascia extraperitonealis) will be applied in the supine position, while posterior release techniques (targeting fascia thoracolumbalis and erector spinae) will be applied in the prone position.
  Arms: Myofascial Release Technique Group
Other: Kinesio Taping Technique — Two different techniques will be used in the Kinesio Taping application. First, four I-shaped Kinesio tapes (Kinesio Tex® Gold), each 5 cm wide and 0.5 mm thick, will be applied in a star-shaped pattern using the "space correction technique" with 25-50% tension at the S2-S4 level (sacral region) while the participant will in a seated position. Additionally, to direct the uterus into retroversion during menstruation, a 15 cm long I-shaped tape will be applied to the suprapubic region using the "ligament correction technique" with 100% tension.
  Arms: Kinesio Taping Group

SUMMARY:
Dysmenorrhea is a physiological condition and one of the most common issues experienced during menstruation. This study aims to compare the acute effects of Myofascial Release Technique (MRT) and Kinesio Taping® (KT) on pain severity, fatigue, and menstrual symptom severity in individuals with primary dysmenorrhea (PD).

DETAILED DESCRIPTION:
A total of 45 individuals diagnosed with PD will be randomly assigned to one of three groups: MRT, KT, or control. Pain severity and fatigue will be measured using the Visual Analog Scale (VAS), while menstrual symptom severity will be assessed with the Menstrual Symptom Scale, both prior to and following the interventions. The MRT group will be received MRT for three consecutive days starting from the onset of menstruation, whereas the KT group will be applied KT application for a duration of 72 hours. The control group did not receive any form of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Daignosed with primary dysmenorrhea
* Regular menstruation in the past six months
* Experience menstrual pain ranging between 40-100 mm on the Visual Analog Scale

Exclusion Criteria:

* Diagnosis of secondary dysmenorrhea
* A menstrual cycle length of less than 21 days or more than 35 days
* A history of childbirth or pregnancy
* Use of pharmacological treatments for menstrual pain
* A history of pelvic pathology or pelvic surgery
* The presence of neurological or systemic diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Pain Severity | 3 months
  A 100 mm Visual Analog Scale (VAS), represented as a straight line with one end marked as 0 (no pain) and the other end as 10 (unbearable pain), will be used to measure pain severity. Participants will be asked to mark the point on the line that corresponded to the level of pain they will be experiencing during the evaluation. The marked point will be then measured using a ruler, and the numerical value of the pain severity will be recorded. Higher results indicate worse pain intensity.
Fatigue | 3 months
  A 100 mm Visual Analog Scale (VAS), with one end marked as 0 (no fatigue) and the other end as 10 (unbearable fatigue), will be used to evaluate the severity of fatigue experienced on the most intense day of menstruation. Participants will be asked to mark the point on the VAS that corresponded to the level of fatigue they will be felt. The marked point will then measured using a ruler, and the numerical value will be recorded. Higher results indicate worse pain intensity.
Menstrual Symptoms | 3 months
  The "Menstrual Symptom Scale," developed by Chesney and Tatso, will be used to evaluate the severity of menstrual symptoms. This scale consists of 22 items, each with five response options, and includes three subdimensions. The first 13 items belong to the "Negative Effects/Somatic Complaints" subdimension, items 14 to 19 fall under the "Menstrual Pain Symptoms" subdimension, and the last three items are part of the "Coping Methods" subdimension. The responses will be rated on a Likert-type scale ranging from 1 (never) to 5 (always). A higher total score indicates greater severity of menstrual symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Miçooğulları, PhD, Principal Investigator — Cyprus International University
Locations (2):
- Turkey (Türkiye) (2):
  - Cyprus International University, Mersin, Haspolat
  - Cyprus International University, Mersin, Lefkosa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma YX, Ma LX, Liu XL, Ma YX, Lv K, Wang D, Liu JP, Xing JM, Cao HJ, Gao SZ, Zhu J. A comparative study on the immediate effects of electroacupuncture at Sanyinjiao (SP6), Xuanzhong (GB39) and a non-meridian point, on menstrual pain and uterine arterial blood flow, in primary dysmenorrhea patients. Pain Med. 2010 Oct;11(10):1564-75. doi: 10.1111/j.1526-4637.2010.00949.x. Epub 2010 Sep 7. PMID 21199306
- [Result] Kaur, A., Ray, G., & Mitra, M. (2017). Comparing the effectiveness of connective tissue mobilisation and kinesio-taping on females with primary dysmenorrhea. Indian Journal of Physiotherapy & Occupational Therapy, 11, 70-5.
- [Result] Harel Z. Dysmenorrhea in adolescents and young adults: etiology and management. J Pediatr Adolesc Gynecol. 2006 Dec;19(6):363-71. doi: 10.1016/j.jpag.2006.09.001. PMID 17174824
- [Result] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680
- [Result] Ajimsha MS. Effectiveness of direct vs indirect technique myofascial release in the management of tension-type headache. J Bodyw Mov Ther. 2011 Oct;15(4):431-5. doi: 10.1016/j.jbmt.2011.01.021. Epub 2011 Feb 11. PMID 21943616